CLINICAL TRIAL: NCT03692468
Title: A Brief Intervention for Co-occurring Pain and Distress in Primary Care
Brief Title: A Brief Intervention for Chronic Pain in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Lisa Matero, Senior Staff Psychologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pain in Primary Care
Record Dates: First submitted 2018-09-20; First posted 2018-10-02 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will engage in a 5 session psychotherapy intervention focused on improving pain and mood.
  Interventions: Behavioral: Psychotherapy
- Control Group (No Intervention): Patients will receive treatment as usual from their care providers.

INTERVENTIONS:
Behavioral: Psychotherapy — Participants will complete 5, 60 minutes sessions. At each session, participants will learn strategies that have been shown to improve pain functioning and/or mood for patients who have chronic pain. The intervention will be delivered in the patient's primary care clinic.
  Arms: Intervention Group

SUMMARY:
The purpose of this research study is to investigate potential benefits of a behavioral intervention for co-occurring chronic pain and distress that is delivered in a primary care clinic.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain condition
* A current patient within the Henry Ford Health System Academic Internal Medicine Clinic in Detroit
* Has been within the Henry Ford Health System for at least 6 months

Exclusion Criteria:

* Current behavioral health treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | 5 weeks post-baseline
  The Brief Pain Inventory measures pain severity and pain functioning. Pain severity is comprised of 4 questions on a 0-10 scale for pain at it's worst in the past week, the least in the past week, on average, and then currently. Each item is scored separately and higher scores indicate greater pain severity. There are then 12 daily activities in which the participants rates on a scale of 0-10 regarding how much the pain interferes with the activity (10 being the highest interference). These are all scored separately.
Hospital Anxiety and Depression Scale | 5 weeks post-baseline
  This measure assesses the severity of depression and anxiety. Scores on each of the subscale (e.g., depression and anxiety) range from 0-21 with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Insomnia Severity Index | Administered at baseline, 5 weeks post-baseline, and 1 month and 6-month follow-ups
  This measure assess difficulty with sleep. Total scores range from 0-28, with greater numbers indicating greater sleep difficulty.
Pain Catastrophizing Scale | Administered at baseline, 5 weeks post-baseline, and 1 month and 6-month follow-ups
  This measure assesses catastrophizing thoughts about pain. Total scores range from 0-52 with higher scores indicating greater catastrophizing. The three subscales are rumination (range= 0-16), magnification (range= 0-12), and helplessness (range= 0-24).
Satisfaction with Life Scale | Administered at baseline, 5 weeks post-baseline, and 1 month and 6-month follow-ups
  This measure assesses how satisfied a patient is with their life. Total scores range from 7-35 with higher scores indicating greater satisfaction.
Health care utilization | Measured 6 months before and 6 months after study enrollment
  The number of primary and specialty care visits, prescriptions written, emergency room visits, and hospital admissions

OTHER OUTCOMES:
Chronic Pain Acceptance Questionnaire | Administered at baseline, 5 weeks post-baseline, and 1 month and 6-month follow-ups
  This measure assess acceptance of chronic pain. Total scores range from 0-120 with higher scores indicating greater acceptance. There are 2 subscales: Activity Engagement (range= 0-66) and Pain Willingness (range= 0-54).
Mindful Attention Awareness Scale | Administered at baseline, 5 weeks post-baseline, and 1 month and 6-month follow-ups
  This measure assess the extent to which someone is using mindful awareness. Total scores range from 15-90 with greater scores indicating greater mindfulness.
Montreal Cognitive Assessment | Administered at baseline
  Brief screen of cognitive functioning; scores range from 0-30
Brief Medical Numbers Test | Administered at baseline
  Brief screen of health numeracy; scores range from 0-4
Rapid Estimate of Adult Learning in Medicine | Administered at baseline
  Brief screen of health literacy; patients are categorized into a reading level: at least 9th grade, 7th-8th grade, 4th-6th grade, and 3rd grade or less

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Derived] Miller-Matero LR, Gavrilova L, Hecht LM, Autio K, Tobin ET, Braciszewski JM, Maye M, Felton JW, Ahmedani BK. A brief psychological intervention for chronic pain in primary care: Examining long-term effects from a pilot randomized clinical trial. Pain Pract. 2022 Jul;22(6):564-570. doi: 10.1111/papr.13134. Epub 2022 Jun 14. PMID 35665994
- [Derived] Miller-Matero LR, Hecht LM, Miller MK, Autio K, Pester BD, Tobin ET, Patel S, Braciszewski JM, Maye M, Ahmedani BK. A Brief Psychological Intervention for Chronic Pain in Primary Care: A Pilot Randomized Controlled Trial. Pain Med. 2021 Jul 25;22(7):1603-1611. doi: 10.1093/pm/pnaa444. PMID 33616190